CLINICAL TRIAL: NCT06110936
Title: Effects of Transcutaneous Spinal Direct Current Stimulation on Mobility in Cases With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Gulser CINBAZ, research assistant, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.2021.733
Record Dates: First submitted 2023-10-23; First posted 2023-11-01 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ts-DCS Group (Experimental): ts-DCS will be administered using a direct current stimulator (TCT Research Limited, Hong Kong). 2-mA intensity ts-DCS will be applied to the experimental group, with the active electrode being the cathode electrode. The two electrodes (35-cm2) to be used will be immersed in saline solution (0.9% NaCl). The stimulation electrode (cathodal) will be placed slightly above the spinous process of the T10 vertebral process, while the reference electrode (anodal) will be placed horizontally on the left deltoid.
  Interventions: Device: Transcutaneous Spinal Direct Current Stimulation
- Control Group (Sham Comparator): ts-DCS will be administered using a direct current stimulator (TCT Research Limited, Hong Kong). 2-mA intensity ts-DCS will be applied to the control group, with the active electrode being the cathode electrode. The two electrodes (35-cm2) to be used will be immersed in saline solution (0.9% NaCl). The stimulation electrode (cathodal) will be placed slightly above the spinous process of the T10 vertebral process, while the reference electrode (anodal) will be placed horizontally on the left deltoid. In the application to the control group, the placement of the electrodes will be the same as the active protocol, and unlike the experimental group, the stimulation will be stopped after 30 seconds. This sham procedure has been reported to be a good pseudostimulation method that does not cause significant experimental effects due to the initial itching sensation it provides.
  Interventions: Device: Transcutaneous Spinal Direct Current Stimulation

INTERVENTIONS:
Device: Transcutaneous Spinal Direct Current Stimulation — Transcutaneous spinal direct current stimulation (ts-DCS), a neuromodulation technique, is one of the non-invasive brain stimulation techniques. ts-DCS occurs when a continuous and low-intensity electric current passes through electrodes with moist sponges placed on the spinal cord.
  Other Names: transvertebral direct current stimulation

SUMMARY:
The primer aim of the study is to examine the effects of the transcutaneous spinal direct current stimulation (ts-DCS) on mobility in addition to the physiotherapy program to individuals with multiple sclerosis. Our secondary aim is to show the relationship of these effects with ts-DCS through fatigue and quality of life evaluations.

DETAILED DESCRIPTION:
Our study is carried out at Istanbul Cadde Medical Center. The patients who will participate in the study are determined according to the inclusion criteria among the patients who applied to the Multiple Sclerosis Polyclinic of Istanbul Medeniyet University Göztepe Training and Research Hospital, Department of Neurology. Transcutaneous spinal direct current will be applied to the individuals participating in our study in 20-minute sessions, 3 days a week for 2 weeks. According to the type of stimulation applied, participants are divided into two groups: experimental and control groups by simple randomization. While cathodal ts-DAU was applied to the patients in the experimental group; Sham ts-DAU is applied to patients in the control group. The same evaluations will be applied to all participants throughout the study, and the evaluations are applied before and after the intervention. The data collected as a result of the evaluations will be analyzed with SPSS version 22.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with MS and suffering from walking difficulties due to MS
* EDSS score between 2-6
* Being over 18 years old

Exclusion Criteria:

* Relapsed within the last two months
* Changed medication within 45 days
* Hospitalized in the last three months
* Had other neurological or musculoskeletal problems
* Had an obstacle to stimulation (skin problems, metal implants, etc.)
* Do not want to participate in the study individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Timed 25-Foot Walk (T25-FW) | It will be evaluated twice: immediately before and immediately after 2 weeks treatment.
  Timed 25 Foot Walking Test was used for objective evaluation of walking. In T25-FW, which evaluates lower extremity function, the individual is asked to walk 25 steps as quickly and safely as possible (if he/she uses a walking aid, this is done together). The time spent walking is recorded in seconds.
Time Up and Go (TUG) | It will be evaluated twice: immediately before and immediately after 2 weeks treatment.
  It is a performance-based test used to evaluate functional mobility and walking speed. The person is asked to get up from the chair he/she is sitting on without support from his/her arms, walk 3 meters at a safe and normal speed, turn around, walk back, sit on the chair again, and the time is recorded in seconds (sec). The test is started with the patient's feet flat on the floor and arms resting on the armrest of the chair. Three repetitions are made and the best result is recorded.
Multiple Sclerosis Walking Scale-12 (MSWS-12) | It will be evaluated twice:immediately before and immediately after 2 weeks treatment.
  It is a 12-item rating scale used to assess individuals' perspectives on the impact of their disease on their ability to walk. During the test, patients are asked to rate how much MS affects their mobility, such as standing, walking, running, and climbing stairs, on a 5-point Likert Scale (1=almost not at all, 5=extremely). A high score indicates that walking ability is affected or the patient has difficulty walking. The lowest score can be 12 and the highest score can be 60 from the test.
Gait Speed Assessment | It will be evaluated twice: immediately before and immediately after 2 weeks treatment.
  Calculation of walking speed will be done by 2D video analysis method. Kinovea 2D motion analysis software (GPLv2 license, 2019) will be used for analysis. The method has validity and reliability. The videos taken with the cameras placed laterally will be uploaded to the program and the necessary calculations will be made.

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) | It will be evaluated twice: immediately before and immediately after 2 weeks treatment.
  The scale, which includes the experience of fatigue, its causes and its effects on daily life, consists of 9 questions and is a Likert-type scale where each question takes a value between 0 and 7. The highest score reached is 63. A score of 36 or above indicates a high perception of fatigue severity.
Fatigue Impact Scale (FIS) | It will be evaluated twice: immediately before and immediately after 2 weeks treatment.
  Fatigue Impact Scale will be used to evaluate the reflection of fatigue on daily activities in patients. This scale evaluates the physical, cognitive and social effects of fatigue in the last month with a total of 40 questions (0 = no problem, 4 = extreme). The total score ranges from 0-160, with higher scores indicating a higher degree of fatigue impact

CONTACTS AND LOCATIONS:
Locations (1):
- Cadde Tıp Merkezi, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No